CLINICAL TRIAL: NCT07154212
Title: Managing the Risk of Hepatitis B Virus Reactivation in COVID-19 Patients Treated With Corticosteroids
Brief Title: Hepatitis B Virus Reactivation in COVID-19
Acronym: HBV-C19
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: HBV in covid
Record Dates: First submitted 2025-09-02; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: COVID-19 Pneumonia; Hypoxemia; Hepatitis B
MeSH Terms: conditions — Hypoxia; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hepatitis B virus infected patients receiving corticosteroids for COVID-19 pneumonia
  Interventions: Diagnostic Test: Hepatitis B virus infection

INTERVENTIONS:
Diagnostic Test: Hepatitis B virus infection — anti-hepatitis B virus core antigen positive serologic status

SUMMARY:
The aim of this observational cohort study was to evaluate adherence to hepatitis B virus (HBV) screening guidelines in a country characterized by low HBV prevalence and assess the potential reactivation and progression of HBV infection in anti-HBV core antigen antibodies (anti-HBc) positive patients receiving corticosteroids for coronavirus disease 2019 (COVID-19).

ELIGIBILITY:
Inclusion Criteria:

* hospitalized adult patients with a positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) ribonucleic acid (RNA) polymerase chain reaction (PCR) test
* supplemental oxygen
* treated with corticosteroids for COVID-19 pneumonia

Exclusion Criteria:

* age under 18 years
* hospitalized for medical conditions unrelated to COVID-19
* received corticosteroid therapy for non-COVID-19 reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized and treated with corticosteroids for covid-19
Sampling Method: Non-Probability Sample
Enrollment: 1793 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
HBV reactivation | at least 3 months post treatment with corticosteroids
  number (%) of patients with HBV reactivation
number (%) of patients with HBV reactivation | one year

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
All anonymous data generated or analyzed during this study are available from the corresponding author upon reasonable request.